CLINICAL TRIAL: NCT00382564
Title: Magnetic Resonance Angiography (MRA) in the Diagnosis of Atherosclerotic Disease Using High Field (3T) MRI Scanners: A Pilot Technical Development Study
Brief Title: Magnetic Resonance Angiography to Diagnose Atherosclerotic Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060249; 06-DK-0249
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2012-05-01

CONDITIONS: Atherosclerosis; Hyperlipidemia; Hypertension; Diabetes Mellitus
Keywords: Imaging; Arteriosclerosis; Hardening of the arteries; MRA; Narrowing of Vessels; Noninvasive Plaque Imaging; Atherosclerotic Disease; Plaque; Arteries; Diabetes; Hypertension
MeSH Terms: conditions — Atherosclerosis; Hyperlipidemias; Hypertension; Diabetes Mellitus; Arteriosclerosis; Plaque, Amyloid

SUMMARY:
This study will determine the usefulness of magnetic resonance imaging (MRI) for examining the heart or blood vessels. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. The subject lies on a table that can slide in and out of the scanner (a metal cylinder), wearing earplugs to muffle loud noises that occur during the scanning process. MRI of the heart and blood vessels, called magnetic resonance angiography (MRA), is a developing diagnostic method that permits evaluation of arteries and veins without the use of x-rays or invasive catheterization required by conventional angiography.

People 18 years of age and older with known or suspected atherosclerotic disease may be eligible for this study.

Participants have blood tests and MRA scanning. The MRA takes about 1.5 to 2 hours. During part of the scan, a contrast agent may be injected into a vein to brighten the images of the heart and blood vessels. Subjects are monitored with an electrocardiogram and are asked to hold their breath for about 5 to 20 seconds intermittently during the procedure.

A CT scan may be done to confirm the MRA findings. CT uses x-rays to produce pictures of the heart and blood vessels. The subject lies on a bed during the scan and is given a contrast agent through a catheter inserted into a vein. Subjects are asked to hold their breath intermittently for about 5 to 20 seconds. A medicine called a beta blocker may be administered to slow the heart rate.

DETAILED DESCRIPTION:
Magnetic Resonance Angiography (MRA) is a developing technique that permits the non-invasive evaluation of arterial and venous structures without the need for x-ray based catheter angiography. While dramatic progress has been made in the last few years, there are still substantial limitations in the accuracy of MRA in the evaluation of coronary artery. The primary aim of this study is to evaluate state-of-the-art techniques for coronary MRA in subjects with known or suspected coronary atherosclerosis. The secondary aim of this protocol is to generate natural history data for future hypothesis-driven clinical trials using MRA techniques developed in this current protocol. The long-term objective of this pilot study and research initiative is to improve coronary MRA to the point that it can reliably replace diagnostic x-ray catheter angiography in the evaluation of subjects with atherosclerotic disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subjects with known or suspected atherosclerotic disease based on clinical findings or documented by angiography (conventional, CT or MRA), or Doppler ultrasound. Subjects at risk for atherosclerosis including: smoking, hyperlipidemia, low levels of high density lipoproteins (less than 50 mg/dl for women and less than 40 mg/dl for men), hypertension, family history (early onset atherosclerosis less than 55 year old in male and less than 65 year old in female who is first degree relative), and diabetes mellitus or metabolic syndrome.
  2. Subject must be willing to participate in the protocol.
  3. Subject age greater than 18 years old.
  4. Subject must be clinically stable and be able to come to the Clinical Center to participate in the study.

EXCLUSION CRITERIA:

1. Subjects with contraindication to MRI scanning. These contraindications include but are not limited to the following devices or conditions:

   1. Implanted cardiac pacemaker or defibrillator
   2. Cochlear Implants
   3. Ocular foreign body (e.g. metal shavings)
   4. Embedded shrapnel fragments
   5. Central nervous system aneurysm clips
   6. Implanted neural stimulator
   7. Medical infusion pumps
   8. Any implanted device that is incompatible with MRI.
2. Unsatisfactory performance status as judged by the referring physician such that the subject could not tolerate an MRI scan. Examples of medical conditions that would not be accepted would include unstable angina and dyspnea at rest.
3. Subjects requiring sedation for MRI studies.
4. Subjects with a condition precluding entry into the scanner (e.g. morbid obesity, claustrophobia, etc.).
5. Pregnant or lactating women.
6. Subjects with severe back-pain or motion disorders who will be unable to tolerate supine positioning within the MRI scanner and hold still for the duration of the examination.
7. Subjects who are unable to undergo a CTA within 1 month of the MRA part of this study, or are unable undergo or be scheduled for a cardiac catheterization within 1 month of the MRA.

   FOR GADOLINIUM BASED MRI STUDIES ONLY:
8. History of severe allergic reaction to gadolinium contrast agents despite the use of premeditation with an anti-histaminic and cortisone.
9. Creatinine value greater than 3.0 mg/dl

   FOR CARDIAC CT:
10. Recent cardiac CT within a month. Both a coronary CTA and calcium score scan are required for this study. If any of these scans were performed at an outside facility and meet the necessary quality level, then that aspect of the cardiac CT scan (coronary CTA, calcium score scan or both) will not be performed at the NIH. Coronary CTA and/or calcium score CT obtained at the outside facility must be performed within one month of subject inclusion and acquired using a 16 slice scanner or higher and should be of good quality. The unformatted images of outside cardiac scans must be available to the primary investigator within one month of their acquisition for eligibility of inclusion in the study.

    FOR CORONARY CTA:
11. Contraindication to the use of CT contrast agents:

    1. Creatinine value greater than 1.4 mg/dl
    2. History of multiple myeloma
    3. Use of metformin-containing products less than 24 hrs prior to contrast administration
    4. History of significant allergic reaction to CT contrast agents despite the use of premeditation with an anti-histaminic and cortisone.
12. Subjects with contraindication precluding the use of beta blockers necessary to perform the coronary CTA. These include:

    1. Asthma
    2. Active bronchospasm
    3. Moderate or severe COPD
    4. Second or third degree AV block
    5. Decompensated cardiac failure
    6. Allergy to beta blockers
    7. Systolic blood pressure less than 100 mm Hg
    8. Pregnancy or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2006-09-25; Study Completion 2012-05-01

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Gharib, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kim WY, Danias PG, Stuber M, Flamm SD, Plein S, Nagel E, Langerak SE, Weber OM, Pedersen EM, Schmidt M, Botnar RM, Manning WJ. Coronary magnetic resonance angiography for the detection of coronary stenoses. N Engl J Med. 2001 Dec 27;345(26):1863-9. doi: 10.1056/NEJMoa010866. PMID 11756576
- [Background] Lopez AD, Murray CC. The global burden of disease, 1990-2020. Nat Med. 1998 Nov;4(11):1241-3. doi: 10.1038/3218. No abstract available. PMID 9809543
- [Background] Hoffmann MH, Shi H, Schmitz BL, Schmid FT, Lieberknecht M, Schulze R, Ludwig B, Kroschel U, Jahnke N, Haerer W, Brambs HJ, Aschoff AJ. Noninvasive coronary angiography with multislice computed tomography. JAMA. 2005 May 25;293(20):2471-8. doi: 10.1001/jama.293.20.2471. PMID 15914747